CLINICAL TRIAL: NCT05368701
Title: Randomised Controlled Trial of a Smartphone-based App to Reduce Self-harm for CAMHS-treated Adolescents
Brief Title: Developing a Smartphone-based App to Reduce Self-harm for CAMHS-treated Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Jessica Leather, Research Associate, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 313791
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Self-harm
Keywords: self-harm; suicidal ideation; suicide attempt; smartphone app; volitional help sheet; implementation intentions; if-then plans
MeSH Terms: conditions — Self-Injurious Behavior; Suicidal Ideation; Suicide, Attempted

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to one of three conditions. Patients will be randomised to the control group or the interventions in a 1:1:1 using a computer-generated random allocation sequence with block sizes of 3, 6, and 9.
Who Masked: Participant, Investigator
Masking Description: The allocation sequence will be concealed from the researcher by using a centralised service (e.g., trial coordination centre) to ensure that selection remains unbiased. Thus, the trial will be double-blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- App-based volitional help sheet (VHS) for self-harm (Experimental): A smartphone-based app version of the adapted VHS for self-harm. Participants read a brief statement designed to encourage them to avoid self-harming ("We want you to plan to avoid self-harming"). Participants are presented with ten 'high risk' situations (temptations). By selecting an appropriate situation, 10 appropriate responses (processes of change) are suggested (see Armitage, 2008). Participants are told that identifying situations in which they were tempted to self-harm and identifying ways to overcome those temptations had been shown to help people change their behaviour.
  Participants in this condition are asked to form implementation intentions by linking critical situations with appropriate responses by choosing an appropriate response from a drop down menu for each critical situation.
  Interventions: Behavioral: Volitional Help Sheet for self-harm
- App-based pencil-and-paper VHS (Active Comparator): The app will deliver a .pdf file (for printing) worksheet of the VHS for self-harm, with no integration into the app.
  Participants read a brief statement designed to encourage them to avoid self-harming ("We want you to plan to avoid self-harming"). Participants are presented with a table with two columns and ten rows. Ten 'high risk' situations (temptations) are presented in the left hand column and 10 appropriate responses (processes of change) are presented in the right hand column (see Armitage, 2008). Participants are told that identifying situations in which they were tempted to self-harm and identifying ways to overcome those temptations had been shown to help people change their behaviour.
  Participants in this condition are asked to form implementation intentions by linking critical situations with appropriate responses by choosing an appropriate response by drawing a line between the situation and response.
  Interventions: Behavioral: Volitional Help Sheet for self-harm
- App with no VHS component (No Intervention): An app with no VHS component that collects questionnaire survey data.
  In this control condition, the app only contains the survey questions and links to helplines contained in the other two conditions.
  A free text entry box will ask participants to think of important situations where they might self-harm. A second box asks participants to think of alternative plans that they can do instead of self-harming. Participants are not guided to make links between the situations and responses.

INTERVENTIONS:
Behavioral: Volitional Help Sheet for self-harm — The "volitional help sheet" (VHS) is a brief psychosocial intervention that significantly reduces thoughts and acts of self-harm in adults admitted to hospital following an initial episode of self-harm. It is based on IF-THEN statements that help people link critical situations to alternative appropriate responses. An example is: "If I feel the urge to self-harm when I want to get relief from a terrible state of mind, then I will do something else instead of self-harming". IF-THEN statements are intended to act as automatic coping responses, especially in cases where people may feel the urge to self-harm.
  The VHS has previously been successful in reducing self-harm in people recently admitted to hospital for self-harm. Recent data have also demonstrated that a web-based version of the VHS was acceptable among a large representative sample of UK adults with self-harm experiences. However, it is yet to be known whether this intervention is effective and acceptable among adolescents.
  Other Names: If-Then Plans
  Arms: App-based pencil-and-paper VHS; App-based volitional help sheet (VHS) for self-harm

SUMMARY:
The aim of the present research is to explore whether a brief, smartphone app-based intervention based on psychological theory can help adolescents to avoid self-harming.

The smartphone app will be piloted in a randomised controlled trial (RCT) with adolescents. 90 adolescents will be recruited and assigned to one of three conditions: (a) intervention group who will complete the smartphone-based VHS app for self-harm (n = 30), (b) control group (n = 30) who will complete paper-and-pencil modified VHS, without the app, and (c) control group who will complete measures via the app but not the VHS (n = 30).

DETAILED DESCRIPTION:
Background Self-harm among young people is frequent (McManus et al., 2019) and presents a growing public health concern in England. To date, no robust and comprehensive evidence base exists for effective interventions to prevent self-harm in adolescents (Witt et al., 2021). Therapeutic interventions that are effective among adults, including dialectical behavioural therapy, are only offered to CAMHS patients being diagnosed with a severe mental illness. Young patients with experiences of self-harm and their carers need to access interventions quickly to improve clinical care and reduce future harm. Therefore, novel interventions need to be developed, tested, and evaluated for this vulnerable population.

One such potential intervention is the "volitional help sheet" (VHS). The VHS is a brief psychosocial intervention that significantly reduces thoughts and acts of self-harm in adults admitted to hospital following an initial episode of self-harm (O'Connor et al., 2017). It is based on IF-THEN statements that help people link critical situations to alternative appropriate responses (Armitage, 2008; Gollwitzer, 1993). An example is: "If I feel the urge to self-harm when I want to get relief from a terrible state of mind, then I will do something else instead of self-harming". IF-THEN statements are intended to act as automatic coping responses, especially in cases where people may feel the urge to self-harm.

The VHS has previously been successful in reducing self-harm in people recently admitted to hospital for self-harm (Armitage et al., 2016; O'Connor et al., 2017). Recent data have also demonstrated that a web-based version of the VHS was acceptable among a large representative sample of UK adults with self-harm experiences (Keyworth et al., 2021). However, it is yet to be known whether this intervention is effective and acceptable among adolescents. It is important to conduct this research with experts by experience to create an acceptable and effective intervention, particularly since talking about self-harm does not increase risk of self-harm (Biddle et al., 2013; Blades et al., 2018), and can actually be positive experience for patients (Alexander et al., 2018; Dazzi et al., 2014). This research will co-adapt and pilot the VHS intervention in adolescents presented at CAMHS following an initial episode of self-harm. To maximise engagement with the intervention, we plan to develop this as a smartphone app.

Methods Design Pilot randomised controlled trial. Participants Adolescents who have previously harmed themselves. Setting Data collection will take place online. We will recruit both adolescents that are currently under the care of CAMHS, and those who have been discharged back to community care.

Recruitment and sampling A sample of 90 adolescents that have experienced and index episode of self-harm will be recruited through purposive sampling via Salford CAMHS and 42nd Street.

Materials A smartphone-based app version of the VHS will be developed. A pencil-and-paper modified VHS will be used for the active control group. A second version of the app will be developed to capture measures for the passive control group.

A novel questionnaire will be developed to run natively within the app to capture measures of effectiveness. Measures of current ideation and history of self-harm episodes alongside demographic information and potential mechanisms (e.g., capabilities, opportunities and motivations to avoid self-harm (Keyworth et al., 2020)) will be collected at baseline and at 6-months post-intervention.

Self-harm will be assessed with three items taken from the British Psychiatric Morbidity Survey (McManus et al., 2016) measuring non-suicidal self-harm (NSSH), suicidal ideation, and suicide attempts. Potential mechanisms will be captured using four measures: exposure to suicide and mental imagery about death; capabilities, opportunities and motivations; habits; and self-regulation. Questions based around the Theoretical Framework of Acceptability (Sekhon et al., 2017) will capture participant perceptions of the acceptability of the intervention. Uptake of the intervention will be measured at follow-up by measuring the frequencies with which critical situations were encountered and appropriate responses were used.

Procedure Data will be collected at two time points over a period of 6 months: baseline, and at six-month follow-up. Participants will be randomised into one of three conditions, to either receive the modified app-based VHS (intervention group; to make links between situations and solutions), a pencil-and-paper VHS (active control group; to make links between situations and solutions), or an app with no VHS component (passive control; where participants asked to identify situations and solutions, without making explicit links between them).

Participants will firstly be asked to complete a short series of demographic questions via an online questionnaire. This will be collected via an online survey which will be emailed to participants in the pencil-and-paper condition, and will be integrated into the app for conditions 1 and 3. Participants will also be asked about their history of self-harm, and questions to assess any psychological aspects involved in self-harm. To test the effectiveness of the intervention measures of non-suicidal self-harm (NSSH), suicidal ideation, and suicide attempts will be assessed via the app's questionnaire.

Participants in the two VHS conditions will be asked to construct "IF-THEN plans" which aim to support patients to reduce self-harm. After participants have created their "IF-THEN plans" they complete a series of questions about their experiences taking part in the intervention. These questions are to assess the feasibility and acceptability of "IF-THEN" plans in the context of self-harm and to iteratively modify the existing VHS. All questions will be optional and participants can choose to skip any should they desire.

Participants in the passive control condition will be asked to identify important situations and coping strategies that they can employ, but without making explicit links.

Ethical considerations Participants will be informed about the study before they agree to take part in it, they are under no obligation to participate in the study, and are free to withdraw from the study at any time, without giving a reason (this information will be in the participant information sheet).

People who self-harm are a vulnerable group who are likely to be experiencing emotional turmoil but they are an essential group to include in research, especially on self-harm services which are of variable quality. Participants may be become emotional when discussing experience with mental health services. However, evidence suggests that participating in research studies can be beneficial for vulnerable groups (Batterham et al., 2018; Blades et al., 2018), and that exposure to suicidal related content does not increase risk of suicidal ideation or engaging in suicidal behaviour (Alexander et al., 2018; Smith et al., 2010).

Our experience running a previous trial using a similar intervention confirms that adverse events are rare. However, there is a low risk of some participants finding the VHS difficult as it may induce uncomfortable emotions or result in distress. This is largely because it focuses on participants identifying situations where they may be tempted to self-harm.

Similarly, our experience running a previous trial using a similar intervention confirms that adverse events are rare, but discussions about inpatient discharge may induce distress.

All participants will be informed of the possible risk of distress in the Participant Information Sheet. Full contact details of the lead researchers will also be provided should participants wish to contact the research team to discuss any queries before they are asked to consent to take part. It will also be suggested to participants that if they feel that taking part in the study induces significant emotional distress or increases feelings related to self-harm, then they may need to reconsider their decision to partake.

All participants will be informed they do not need to answer any questions they do not wish to. They also will be free to withdraw from the study at any time without any penalties. Participants will be advised to withdraw from the study at any point should they become distressed (possibly stopping altogether or taking a break depending on how the participant wants to proceed). Where participants experience significant distress, they will be encouraged to speak with their GP about this at the earliest opportunity.

Participants will have a history of self-harm and it is possible that participants will engage in self-harm during or following the study. Therefore, there may be instances where confidentiality needs to be broken (e.g.: reports of self-harm). Participants will be made fully aware of the limits of confidentiality via the information sheet and consent form. A list of self-harm resources will also be provided as part of the participant Information Sheet.

Participants can opt out of the survey at any time if they are experiencing distress. A page with contact information for support services (e.g., NHS 111, MIND, the Samaritans, Saneline) will be included in the survey for any patients who may become distressed while discussing the subject matter in the online survey.

Researchers will have experience of working on sensitive topics and will meet regularly with the wider research team where any concerns can be reflected upon and discussed.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged between 12-18, who have been admitted to acute mental health in the past year or diagnosed with functional mental health problems

Exclusion Criteria:

* Individuals who cannot give informed consent, or whose parent/guardian cannot give informed consent.
* Individuals under the age of 12 years

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Non-suicidal self-harm | 6 months
  'Have you ever deliberately harmed yourself in any way but not with the intention of killing yourself? (i.e., self-harm)' (British Psychiatric Morbidity Survey) Response option is 'Yes' or 'No'. If respondents answer yes, timing of last episode and frequency will be asked.
Suicidal ideation | 6 months
  'Have you ever seriously thought of taking your life, but not actually attempted to do so?' (British Psychiatric Morbidity Survey) Response option is 'Yes' or 'No'. If respondents answer yes, timing of last episode and frequency will be asked.
Suicide attempt | 6 months
  'Have you ever made an attempt to take your life, by taking an overdose of tablets or in some other way?' (British Psychiatric Morbidity Survey) Response option is 'Yes' or 'No'. If respondents answer yes, timing of last episode and frequency will be asked.

SECONDARY OUTCOMES:
Exposure to suicide and mental imagery about death | 6 months
  Measured at baseline and follow-up using seven items adapted from those used in the literature previously (https://pubmed.ncbi.nlm.nih.gov/26247914/). Calculated as a binary variable ('yes' or 'no). Exposure to mental imagery will be calculated as a total score.
Capability, opportunity and motivation (based on Capability, Opportunity, Motivation-Behaviour model) | 6 months
  Measured using the Capability, Opportunity, Motivation questionnaire (https://pubmed.ncbi.nlm.nih.gov/32314500/). Each of the items (0-10 scale) will be analysed separately as these each measure a separate construct. Higher scores indicate higher agreement with statements.
Habit | 6 months
  Measured using the self-reported habit index (automaticity scale; https://ijbnpa.biomedcentral.com/articles/10.1186/1479-5868-9-102). This consists of four items (each from 1 to 7). Items are scored from 1 to 7, with a higher mean score indicating higher agreement with the statements.
State self-regulation | 6 months
  Items are adapted from those used previously (https://www.tandfonline.com/doi/abs/10.1080/08870440512331317670).
  Mean of the two items for each of three sub-constructs: awareness of standards, self-monitoring, and self-regulatory effort. Items are scored from 1 to 7, with higher scores indicating higher agreement with the statements.
Frequencies with which critical situations were encountered and appropriate responses were used | 6 months
  Frequencies

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Armitage, Principal Investigator — University of Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexander S, Pillay R, Smith B. A systematic review of the experiences of vulnerable people participating in research on sensitive topics. Int J Nurs Stud. 2018 Dec;88:85-96. doi: 10.1016/j.ijnurstu.2018.08.013. Epub 2018 Sep 3. PMID 30219697
- [Background] Armitage CJ. A volitional help sheet to encourage smoking cessation: a randomized exploratory trial. Health Psychol. 2008 Sep;27(5):557-66. doi: 10.1037/0278-6133.27.5.557. PMID 18823182
- [Background] Armitage CJ, Rahim WA, Rowe R, O'Connor RC. An exploratory randomised trial of a simple, brief psychological intervention to reduce subsequent suicidal ideation and behaviour in patients admitted to hospital for self-harm. Br J Psychiatry. 2016 May;208(5):470-6. doi: 10.1192/bjp.bp.114.162495. Epub 2016 Jan 7. PMID 26743808
- [Background] Batterham PJ, Calear AL, Carragher N, Sunderland M. Prevalence and predictors of distress associated with completion of an online survey assessing mental health and suicidality in the community. Psychiatry Res. 2018 Apr;262:348-350. doi: 10.1016/j.psychres.2017.08.048. Epub 2017 Aug 23. PMID 28843625
- [Background] Biddle L, Cooper J, Owen-Smith A, Klineberg E, Bennewith O, Hawton K, Kapur N, Donovan J, Gunnell D. Qualitative interviewing with vulnerable populations: individuals' experiences of participating in suicide and self-harm based research. J Affect Disord. 2013 Mar 5;145(3):356-62. doi: 10.1016/j.jad.2012.08.024. Epub 2012 Sep 25. PMID 23021191
- [Background] Blades CA, Stritzke WGK, Page AC, Brown JD. The benefits and risks of asking research participants about suicide: A meta-analysis of the impact of exposure to suicide-related content. Clin Psychol Rev. 2018 Aug;64:1-12. doi: 10.1016/j.cpr.2018.07.001. Epub 2018 Jul 5. PMID 30014862
- [Background] Dazzi T, Gribble R, Wessely S, Fear NT. Does asking about suicide and related behaviours induce suicidal ideation? What is the evidence? Psychol Med. 2014 Dec;44(16):3361-3. doi: 10.1017/S0033291714001299. Epub 2014 Jul 7. PMID 24998511
- [Background] Keyworth C, Epton T, Goldthorpe J, Calam R, Armitage CJ. Acceptability, reliability, and validity of a brief measure of capabilities, opportunities, and motivations ("COM-B"). Br J Health Psychol. 2020 Sep;25(3):474-501. doi: 10.1111/bjhp.12417. Epub 2020 Apr 20. PMID 32314500
- [Background] Keyworth C, O'Connor R, Quinlivan L, Armitage CJ. Acceptability of a Brief Web-Based Theory-Based Intervention to Prevent and Reduce Self-harm: Mixed Methods Evaluation. J Med Internet Res. 2021 Sep 14;23(9):e28349. doi: 10.2196/28349. PMID 34518153
- [Background] McManus S, Gunnell D, Cooper C, Bebbington PE, Howard LM, Brugha T, Jenkins R, Hassiotis A, Weich S, Appleby L. Prevalence of non-suicidal self-harm and service contact in England, 2000-14: repeated cross-sectional surveys of the general population. Lancet Psychiatry. 2019 Jul;6(7):573-581. doi: 10.1016/S2215-0366(19)30188-9. Epub 2019 Jun 4. PMID 31175059
- [Background] O'Connor RC, Ferguson E, Scott F, Smyth R, McDaid D, Park AL, Beautrais A, Armitage CJ. A brief psychological intervention to reduce repetition of self-harm in patients admitted to hospital following a suicide attempt: a randomised controlled trial. Lancet Psychiatry. 2017 Jun;4(6):451-460. doi: 10.1016/S2215-0366(17)30129-3. Epub 2017 Apr 20. PMID 28434871
- [Background] Sekhon M, Cartwright M, Francis JJ. Acceptability of healthcare interventions: an overview of reviews and development of a theoretical framework. BMC Health Serv Res. 2017 Jan 26;17(1):88. doi: 10.1186/s12913-017-2031-8. PMID 28126032
- [Background] Cukrowicz K, Smith P, Poindexter E. The effect of participating in suicide research: does participating in a research protocol on suicide and psychiatric symptoms increase suicide ideation and attempts? Suicide Life Threat Behav. 2010 Dec;40(6):535-43. doi: 10.1521/suli.2010.40.6.535. PMID 21198322
- [Background] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Interventions for self-harm in children and adolescents. Cochrane Database Syst Rev. 2021 Mar 7;3(3):CD013667. doi: 10.1002/14651858.CD013667.pub2. PMID 33677832
- See also: Related Info — http://www.statisticsauthority.gov.uk/assessment/code-of-practice